CLINICAL TRIAL: NCT00791791
Title: Evaluation of Surgical Stress Index (SSI) During Sevoflurane/Remifentanil Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Berthold Bein, Prof. Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: SSI-134-1
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Analgesia
Keywords: Anesthesia General; Anesthetics Inhalation; Stress measurement; Surgical Stress; Diagnostic Techniques and Procedures
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): increasing remifentanil administration
  Interventions: Procedure: standardized pain stimulus
- 2 (Other): decreasing remifentanil concentration
  Interventions: Procedure: standardized pain stimulus

INTERVENTIONS:
Procedure: standardized pain stimulus — a tetanic stimulus (30s, 50 Hz, 60mA) applied as standardized pain stimulus

SUMMARY:
The aim of the present prospective randomized study was to challenge the ability of SSI to detect painful stimulation during sevoflurane - remifentanil anesthesia.

DETAILED DESCRIPTION:
General anesthesia can be considered as a combination of hypnosis, antinociception and immobility. Whereas monitoring of depth of hypnosis, and muscle relaxation can be regarded as accepted, determination of the nociception is based on clinical signs like somatic or autonomic responses.

Recently, the multivariate surgical stress index (SSI)has been demonstrated to correlate with surgical stress intensity. Thus, SSI might be a useful variable to adjust analgesic drug administration in individual patients.

We want to investigate whether SSI is able to indicate nociception following standardized noxious stimulation during balanced sevoflurane - remifentanil anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* ASA physical status 1-2
* elective surgery in general anesthesia of 1 to 2 hours
* written informed consent

Exclusion Criteria:

* pregnancy
* history of cardiac arrhythmia
* presence of any neuromuscular or neurological disease
* use of CNS-active medication or abuse of alcohol or illicit drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
SSI, compared to standard monitoring variables | during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Gruenewald, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel; Berthold Bein, MD, DEAA, Study Chair — Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Gruenewald M, Zhou J, Schloemerkemper N, Meybohm P, Weiler N, Tonner PH, Scholz J, Bein B. M-Entropy guidance vs standard practice during propofol-remifentanil anaesthesia: a randomised controlled trial. Anaesthesia. 2007 Dec;62(12):1224-9. doi: 10.1111/j.1365-2044.2007.05252.x. PMID 17991257
- [Background] Rehberg B, Grunewald M, Baars J, Fuegener K, Urban BW, Kox WJ. Monitoring of immobility to noxious stimulation during sevoflurane anesthesia using the spinal H-reflex. Anesthesiology. 2004 Jan;100(1):44-50. doi: 10.1097/00000542-200401000-00011. PMID 14695723
- [Derived] Gruenewald M, Meybohm P, Ilies C, Hocker J, Hanss R, Scholz J, Bein B. Influence of different remifentanil concentrations on the performance of the surgical stress index to detect a standardized painful stimulus during sevoflurane anaesthesia. Br J Anaesth. 2009 Oct;103(4):586-93. doi: 10.1093/bja/aep206. Epub 2009 Jul 31. PMID 19648155